CLINICAL TRIAL: NCT03371173
Title: A Pilot Study to Explore Preliminary Safety, Tolerability and Efficacy of ORal IrON Supplementation With Ferric Maltol in Treating Iron Deficiency in Patients With Pulmonary Hypertension and Iron Deficiency Anemia
Brief Title: ORal IrON Supplementation With Ferric Maltol in Patients With Pulmonary Hypertension (ORION-PH-1)
Acronym: ORION-PH-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment rate; difficulties to achieve planned number of participants within reasonable time frame
Sponsor: Hannover Medical School (Other)
Collaborators: Shields, Shields and Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORION-PH-1
Record Dates: First submitted 2017-10-16; First posted 2017-12-13 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2019-06

CONDITIONS: Hypertension, Pulmonary; Anemia, Iron Deficiency
Keywords: Pulmonary Hypertension; Iron Deficiency
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric maltol

STUDY DESIGN:
Intervention Model Description: Explorative, open-label, uncontrolled monocenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferric maltol 30 mg (Feraccru®) (Experimental): Treatment with Feraccru® 30 mg hard capsules (Ferric maltol 30 mg). One capsule twice daily, morning and evening, on an empty stomach for 12 weeks
  Interventions: Drug: Ferric maltol 30 mg (Feraccru®)

INTERVENTIONS:
Drug: Ferric maltol 30 mg (Feraccru®) — Feraccru® 30 mg hard capsules will be used. Each capsule contains 30 mg iron (as ferric maltol), 91.5 mg of lactose, 0.5 mg of Allura Red AC (E129) and 0.3 mg Sunset Yellow FCF (E110) as excipients with known effects

SUMMARY:
This is an explorative, open-label, uncontrolled, single center study to explore the preliminary safety, tolerability and efficacy of oral ferric maltol in treating iron deficiency in patients with pulmonary hypertension and iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any study-related procedure and willingness to comply with treatment and follow-up procedures
2. Male and female patients ≥18 years at day of inclusion
3. Patients capable of understanding the investigational nature, potential risks and benefits of the clinical trial
4. Patients with a diagnosis of PH confirmed by a (historical) right heart catheterization showing a mean pulmonary artery pressure ≥25 mmHg at rest and stable PH medication for at least 3 months.
5. 6 min walk distance >50 m
6. Mild-to-moderate iron-deficiency anemia as defined by a hemoglobin concentration ≥7 g/dl and <12 g/dl in females or ≥8 g/dl and <13 g/dl in males, and serum ferritin <100 µg/l, or 100-300 µg/l and transferrin saturation <20% at screening
7. Prevention of pregnancy:

Women without childbearing potential defined as follows:

* at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
* hysterectomy or uterine agenesis or
* ≥ 50 years and in postmenopausal state ≥ 1 year or
* < 50 years and in postmenopausal state ≥ 1 year with serum FSH > 40 IU/l and serum oestrogen < 30 ng/l or a negative oestrogen test or

Women of childbearing potential with a negative ß-HCG pregnancy test at screening who agree to meet one of the following criteria from the time of screening, during the study and for a period of four weeks following the last administration of study medication:

* correct use of contraception methods. The following are acceptable: hormonal contraceptives (combined oral contraceptives and oestrogen-free pills with desogestrel, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUS) or a barrier method, e.g. condom or occlusive cap (diaphragm or cervical/vault caps) with spermicide (foam, gel, film, cream or suppository)
* true abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception)
* sexual relationship only with female partners and/or sterile male partners

Exclusion Criteria:

1. Active hematological disorders other than iron-deficiency anemia
2. Other medical condition that according to the investigator's assessment is causing or contributing to anemia
3. Active malignancy
4. Active infectious disease
5. Active bleeding
6. Severe renal insufficiency (glomerular filtration rate <30 ml/min)
7. Severe liver injury as indicated by serum aminotransferases >3 x upper limit of normal or bilirubin levels >50 µmol/l
8. Ongoing oral or intravenous iron supplementation
9. Hemoglobin <7 g/dl in females or <8 g/dl in males at screening
10. Concomitant erythropoietin medication
11. Pregnancy or lactation period
12. Subject has received any investigational medication or any investigational device within 30 days prior to the first dose of study medication or is actively participating in any investigational drug/devices trial, or is scheduled to receive an investigational drug/device during the course of the study.
13. Known or suspected hypersensitivity to any of the active substances or any excipients of the investigational medicinal product
14. Known haemochromatosis or other iron overload syndromes
15. Patients who have been receiving repeated (>1) blood transfusions during the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin level from baseline to week 12 | baseline to week 12
  measurement of hemoglobin in blood

SECONDARY OUTCOMES:
Change in hemoglobin from baseline to week 6 | baseline to week 6
  measurement of hemoglobin in blood
Change in serum ferritin levels from baseline to week 6 and 12 | baseline to week 6 and baseline to week 12
  measurement of serum ferritin levels
Change in transferrin saturation from baseline to week 6 and 12 | baseline to week 6 and baseline to week 12
  measurement of transferrin saturation
Change in 6 min walking distance from baseline to week 12 | baseline to week 12
  measurement of functional exercise capacity
Change in serum NT-proBNP from baseline to weeks 6 and 12 | baseline to week 6 and baseline to week 12
  measurement of serum NT-proBNP
Change in echocardiographic markers of right ventricular function from baseline to week 12 (1) | from baseline to week 12
  measurement of right atrial area
Change in echocardiographic markers of right ventricular function from baseline to week 12 (2) | from baseline to week 12
  measurement of right ventricular diameter
Change in echocardiographic markers of right ventricular function from baseline to week 12 (3) | from baseline to week 12
  measurement of fractional area change
Change in echocardiographic markers of right ventricular function from baseline to week 12 (4) | from baseline to week 12
  measurement of tricuspid annular plane systolic excursion
Change in World Health Organization Functional Class (WHO FC) from baseline to week 6 and week 12 | from baseline to week 6 and week 12
  measurement of different parameter according to an evaluated process

OTHER OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | first application of IMP until 4 weeks after treatment discontinuation
  Number of Adverse Events
Incidence of Serious Adverse Events [Safety and Tolerability] | first application of IMP until 4 weeks after treatment discontinuation
  Number of Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Marius Hoeper, Prof. Dr., Principal Investigator — Hannover Medical School, Department of Pneumology
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Olsson KM, Fuge J, Brod T, Kamp JC, Schmitto J, Kempf T, Bauersachs J, Hoeper MM. Oral iron supplementation with ferric maltol in patients with pulmonary hypertension. Eur Respir J. 2020 Nov 12;56(5):2000616. doi: 10.1183/13993003.00616-2020. Print 2020 Nov. PMID 32444411